CLINICAL TRIAL: NCT01334307
Title: Randomized Controlled Trial Of RePneu (LVRC) Endobronchial Coils For The Treatment Of Severe Emphysema With Hyperinflation (RESET Study)
Brief Title: Randomized Comparison of the RePneu Lung Volume Reduction Coil (LVRC) to Standard of Care for the Treatment of Emphysema (RESET Study)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Collaborators: PneumRx, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CLN0008
Record Dates: First submitted 2011-04-01; First posted 2011-04-13 (Estimated); Last update posted 2021-07-21 (Actual); Status verified 2021-07

CONDITIONS: Emphysema
Keywords: Emphysema; RePneu
MeSH Terms: conditions — Emphysema

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lung Volume Reduction Coil (LVRC) (Experimental): Lung Volume Reduction Coil (LVRC)
  Interventions: Device: Lung Volume Reduction Coil (LVRC) (PneumRx)
- Control (Placebo Comparator): Standard of Care
  Interventions: Device: Control

INTERVENTIONS:
Device: Lung Volume Reduction Coil (LVRC) (PneumRx) — Lung Volume Reduction Coil (LVRC)
  Other Names: LVRD
  Arms: Lung Volume Reduction Coil (LVRC)
Device: Control — Standard of Care
  Other Names: LVRC Control treatment is Standard of Care
  Arms: Control

SUMMARY:
The objective of this study is to demonstrate the safety and performance of the PneumRx, Inc. Lung Volume Reduction Coil (LVRC) in a population of patients with emphysema. The PneumRx, Inc. LVRC is used as a less invasive alternative to lung volume reduction surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patient greater than or equal to 35 years of age
* High resolution CT scan indicates unilateral or bilateral emphysema
* High resolution CT scan indicates homogeneous or heterogeneous emphysema
* Patient has post-bronchodilator FEV1 less than or equal to 45% predicted
* Total Lung Capacity greater than 100% predicted
* Patient has marked dyspnea scoring greater than or equal to 2 on mMRC scale of 0-4
* Patient has stopped smoking for a minimum of 8 weeks prior to entering the study
* Patient (and legal guardian if applicable) read, understood and signed the Informed Consent form

Exclusion Criteria:

* Patient has a change in FEV1 greater than 20% post-bronchodilator
* Patients DLCO less than 20% predicted
* Patient has a history of recurrent clinically significant respiratory infection
* Patient has uncontrolled pulmonary hypertension defined by right ventricular pressure greater than 50mm Hg and/or evidenced by echocardiogram
* Patient has an inability to walk greater than 140 meters (150 yards) in 6 minutes
* Patient has evidence of other disease that may compromise survival such as lung cancer, renal failure, etc
* Patient is pregnant or lactating
* Patient has an inability to tolerate bronchoscopy under heavy sedation or anesthesia
* Patient has clinically significant bronchiectasis
* Patient has giant bullae greater than 1/3 lung volume
* Patient has had previous LVR surgery, lung transplant or lobectomy
* Patient has been involved in other pulmonary drug studies with 30 days prior to this study
* Patient is taking greater than 20 mg prednisone (or similar steroid) daily
* Patient is on Plavix or has not been weaned off prior to procedure
* Patient has other disease that would interfere with completion of study, follow up assessments or that would adversely affect outcomes

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2010-02; Primary Completion 2013-06 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
St. George's Respiratory Questionnaire (SGRQ) | three month Follow-Up Visit
  The primary efficacy endpoint will be the difference between treatment and control groups in the change in St. George's Respiratory Questionnaire (SGRQ) from Baseline (Pre-Treatment Visit) to the three month Follow-Up Visit.

CONTACTS AND LOCATIONS:
Overall Officials: Pallav Shah, MD, Principal Investigator — Chelsea and Westminster Hospital
Locations (3):
- United Kingdom (3):
  - Glasgow
  - Chelsea and Westminster Hospital, London
  - Manchester

REFERENCES:
- [Derived] Zoumot Z, Kemp SV, Singh S, Bicknell SR, McNulty WH, Hopkinson NS, Ross ET, Shah PL. Endobronchial coils for severe emphysema are effective up to 12 months following treatment: medium term and cross-over results from a randomised controlled trial. PLoS One. 2015 Apr 8;10(4):e0122656. doi: 10.1371/journal.pone.0122656. eCollection 2015. PMID 25853697
- [Derived] Shah PL, Zoumot Z, Singh S, Bicknell SR, Ross ET, Quiring J, Hopkinson NS, Kemp SV; RESET trial Study Group. Endobronchial coils for the treatment of severe emphysema with hyperinflation (RESET): a randomised controlled trial. Lancet Respir Med. 2013 May;1(3):233-40. doi: 10.1016/S2213-2600(13)70047-X. Epub 2013 Apr 23. PMID 24429129